CLINICAL TRIAL: NCT07131696
Title: The Effect of Transcutaneous Vagal Nerve Stimulation (tVNS) on Cerebral Vasospasm Secondary to Aneurysmal Subarachnoid Hemorrhage
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marshall Holland (Other)
Responsible Party: Sponsor-Investigator, Marshall Holland, Assistant Professor of Neurosurgery, University of Alabama at Birmingham
Organization: University of Alabama at Birmingham (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300015166
Record Dates: First submitted 2025-07-29; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage; Vasospasm, Cerebral; Transcutaneous Vagal Nerve Stimulation (tVNS); Endovascular Treatment
Keywords: CVS; aSAH; tVNS
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tVNS (Experimental)
  Interventions: Device: Transcutaneous Vagal Nerve Stimulation

INTERVENTIONS:
Device: Transcutaneous Vagal Nerve Stimulation — Participants will receive up to 4 sessions per day of up to 20-minute stimulation, over the next 10 days of their inpatient hospital stay, following endovascular treatment. Stimulation will be provided by the tVNS device through a small electrode placed around the ear that will send low intensity, pulsed, electrical pulses the vagus nerve.
  Other Names: tVNS

SUMMARY:
The significance of developing a safe and effective therapy for aneurysmal subarachnoid hemorrhage (aSAH) patients suffering cerebral vasospasm (CVS) cannot be overstated. Vasospasm - a clamping down of normal arteries in the days following rupture - remains incredibly challenging to treat.1,2 Current drugs and minimally invasive surgical therapies are helpful, yet woefully insufficient. Symptomatic cerebral vasospasm afflicts about 30% of aneurysmal subarachnoid hemorrhage patients and nearly half will go on to suffer a stroke, despite aggressive medical care.1-3 The autonomic nervous system is a balance between sympathetic (fight or flight) and parasympathetic (rest and digest) influence with sympathetic overactivity and inflammation shown to play an important role in the development and severity of cerebral vasospasm.4,5,17-20 Prior studies of autonomic nervous system neuromodulation highlight its promise as a promising potential avenue to improve morbidity and mortality from CVS in aSAH.6-15 Despite progress, continued high levels of CVS morbidity and mortality stress the urgent need for exploration of neuromodulation therapy.

In this proposal, the study team will modulate the autonomic nervous system function in aSAH patients using transcutaneous vagal nerve stimulation (tVNS). tVNS involves placement of a stimulation electrode on the external ear to non-invasively stimulate a branch of the vagal nerve and increase parasympathetic influence. This device has FDA approval for epilepsy and cluster headache.

The study hypothesis is that neuromodulation of the autonomic nervous system with tVNS (increasing parasympathetic influence) reduces sympathetic overactivity and inflammation in aSAH resulting in decreased morbidity of CVS.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or Female
* 18-65 years of age
* Diagnosed with Fisher grade 3 or 4 aneurysmal subarachnoid hemorrhage
* Ability to undergo endovascular treatment of aneurysmal subarachnoid hemorrhage
* For females of reproductive potential: negative pregnancy test at time of treatment.
* Plan to undergo standard of care treatment and follow-up

Exclusion Criteria:

* Medically unfit to undergo endovascular treatment (e.g., Hunt Hess grade 5)
* Does not provide consent
* Posterior circulation aneurysmal subarachnoid hemorrhage
* Initial aneurysm treatment after post bleed day 1

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants affected by cerebral inflammation during the course of the study as assessed by laboratory markers in blood and cerebral spinal fluid | Pre-op, Day 1, 2, 7, 10, and discharge (assessed up to 21 days)
Rate of blood flowing through the brain as assessed by transcranial doppler imaging | Pre-op, Day 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, and discharge (assessed up to 21 days)
Number of participants experiencing sudden health issues during the study as determined by the need for ventriculoperitoneal shunt placement prior to discharge, length of hospital stay, and disposition upon discharge. | Pre-op, Day 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, and discharge (assessed up to 21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Marshall Holland, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Hospital, Birmingham, Alabama, United States

REFERENCES:
- [Background] Mazzone P, Rodriguez G, Arrigo A, Nobili F, Pisani R, Rosadini G. Cerebral haemodynamic changes induced by spinal cord stimulation in man. Ital J Neurol Sci. 1996 Feb;17(1):55-7. doi: 10.1007/BF01995709. PMID 8742988
- [Background] Isono M, Kaga A, Fujiki M, Mori T, Hori S. Effect of spinal cord stimulation on cerebral blood flow in cats. Stereotact Funct Neurosurg. 1995;64(1):40-6. doi: 10.1159/000098732. PMID 8751313
- [Background] Phillips I, Johns MA, Pandza NB, Calloway RC, Karuzis VP, Kuchinsky SE. Three Hundred Hertz Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) Impacts Pupil Size Non-Linearly as a Function of Intensity. Psychophysiology. 2025 Feb;62(2):e70011. doi: 10.1111/psyp.70011. PMID 40013407
- [Background] Tekdemir I, Aslan A, Elhan A. A clinico-anatomic study of the auricular branch of the vagus nerve and Arnold's ear-cough reflex. Surg Radiol Anat. 1998;20(4):253-7. PMID 9787391
- [Background] White JC. Nervous control of the cerebral vascular system. Clin Neurosurg. 1963;9:67-87. doi: 10.1093/neurosurgery/9.cn_suppl_1.67. No abstract available. PMID 4954928
- [Background] Edvinsson L, Uddman R, Juul R. Peptidergic innervation of the cerebral circulation. Role in subarachnoid hemorrhage in man. Neurosurg Rev. 1990;13(4):265-72. doi: 10.1007/BF00346363. PMID 2126362
- [Background] Hara H, Edvinsson L. Perivascular innervation of the cerebral circulation: involvement in the pathophysiology of subarachnoid hemorrhage. Neurosurg Rev. 1987;10(3):171-9. doi: 10.1007/BF01782043. PMID 3332035
- [Background] Slavin KV, Vannemreddy P. Cervical spinal cord stimulation for prevention and treatment of cerebral vasospasm after aneurysmal subarachnoid hemorrhage: clinical and radiographic outcomes of a prospective single-center clinical pilot study. Acta Neurochir (Wien). 2022 Nov;164(11):2927-2937. doi: 10.1007/s00701-022-05325-4. Epub 2022 Aug 3. PMID 35920945
- [Background] Takanashi Y, Shinonaga M. Spinal cord stimulation for cerebral vasospasm as prophylaxis. Neurol Med Chir (Tokyo). 2000 Jul;40(7):352-6; discussion 356-7. doi: 10.2176/nmc.40.352. PMID 10927901
- [Background] Holwerda SW, Holland MT, Reddy CG, Pierce GL. Femoral vascular conductance and peroneal muscle sympathetic nerve activity responses to acute epidural spinal cord stimulation in humans. Exp Physiol. 2018 Jun;103(6):905-915. doi: 10.1113/EP086945. Epub 2018 May 5. PMID 29603444
- [Background] Bombardieri AM, Albers GW, Rodriguez S, Pileggi M, Steinberg GK, Heit JJ. Percutaneous cervical sympathetic block to treat cerebral vasospasm and delayed cerebral ischemia: a review of the evidence. J Neurointerv Surg. 2023 Dec;15(12):1212-1217. doi: 10.1136/jnis-2022-019838. Epub 2022 Dec 6. PMID 36597947
- [Background] Jain V, Rath GP, Dash HH, Bithal PK, Chouhan RS, Suri A. Stellate ganglion block for treatment of cerebral vasospasm in patients with aneurysmal subarachnoid hemorrhage - A preliminary study. J Anaesthesiol Clin Pharmacol. 2011 Oct;27(4):516-21. doi: 10.4103/0970-9185.86598. PMID 22096287
- [Background] Suzuki J, Iwabuchi T, Hori S. Cervical sympathectomy for cerebral vasospasm after aneurysm rupture. Neurol Med Chir (Tokyo). 1975;15 pt 1:41-50. doi: 10.2176/nmc.15pt1.41. No abstract available. PMID 60719
- [Background] Wan H, AlHarbi BM, Macdonald RL. Mechanisms, treatment and prevention of cellular injury and death from delayed events after aneurysmal subarachnoid hemorrhage. Expert Opin Pharmacother. 2014 Feb;15(2):231-43. doi: 10.1517/14656566.2014.865724. Epub 2013 Nov 27. PMID 24283706
- [Background] Baggott CD, Aagaard-Kienitz B. Cerebral vasospasm. Neurosurg Clin N Am. 2014 Jul;25(3):497-528. doi: 10.1016/j.nec.2014.04.008. PMID 24994087
- [Background] Dorsch NW. Cerebral arterial spasm--a clinical review. Br J Neurosurg. 1995;9(3):403-12. doi: 10.1080/02688699550041403. PMID 7546361
- [Background] Dorsch N. A clinical review of cerebral vasospasm and delayed ischaemia following aneurysm rupture. Acta Neurochir Suppl. 2011;110(Pt 1):5-6. doi: 10.1007/978-3-7091-0353-1_1. PMID 21116906